CLINICAL TRIAL: NCT03268473
Title: Effect of Non-surgical Periodontal Treatment on Oxidative Stress and Antioxidant Status in Obstructive Sleep Apnea Syndrome (OSAS)
Brief Title: Effect of Non-surgical Periodontal Treatment on Oxidative Stress and Antioxidant Status in OSAS
Acronym: OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: boz001
Record Dates: First submitted 2017-08-22; First posted 2017-08-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Periodontitis; Obstructive Sleep Apnea; OSAS
Keywords: OSAS; Obstructive Sleep Apnea; Periodontitis
MeSH Terms: conditions — Periodontitis; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: It's an assessor blinded, parallel group, randomized controlled trial aimed at investigate whether non-surgical periodontal treatment on serum and saliva oxidative stress parameters in patients with periodontitis and obstructive sleep apnea syndrome (OSAS) and in patients with periodontitis only.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Non-surgical periodontal therapy in patient with OSAS and Periodontitis (Experimental): Non-surgical periodontal therapy consisted of scaling and root planing and supportive periodontal therapy during 3 months Individuals: with both OSAS and periodontitis Intervention: Procedure: Non-surgical periodontal therapy
  Interventions: Other: Experimental
- Control: non-surgical periodontal therapy in Periodontitis (Active Comparator): Non-surgical periodontal therapy consisted of scaling and root planing and supportive periodontal therapy during 3 months Individuals: only periodontitis Intervention: Procedure: Non-surgical periodontal therapy
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — Experimental: Non-surgical periodontal therapy in patient with OSAS and Periodontitis
  Arms: Experimental: Non-surgical periodontal therapy in patient with OSAS and Periodontitis
Other: Control — Control: Non-surgical periodontal therapy in Periodontitis
  Arms: Control: non-surgical periodontal therapy in Periodontitis

SUMMARY:
The main objective of this study is to compare the effect of the non-surgical periodontal treatment on serum and saliva oxidative stress parameters in patients with periodontitis and obstructive sleep apnea syndrome (OSAS) and in patients with periodontitis only.

DETAILED DESCRIPTION:
There is evidence supporting that OSAS is an independent risk factor for cardiovascular and cerebrovascular diseases such as hypertension, congestive heart failure, myocardial infarction, cardiac-arrhythmia, and stroke.Gender, age, smoking, obesity and diabetes, which are risk factors for periodontitis,It is also common in OSAS at the same time.In addition to common risk factors, both OSAS and periodontitis have been shown to be associated with increased oxidative stress markers.

The investigators aimed to investigate whether non-surgical periodontal treatment on serum and saliva oxidative stress parameters in patients with periodontitis and obstructive sleep apnea syndrome (OSAS) and in patients with periodontitis only.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years old
* having more than 16 teeth
* BMI>25 kg/m2

Exclusion Criteria:

* patients with a history of diabetes mellitus or respiratory diseases
* patients who were under any medication that was known to influence periodontal tissues
* patients with a history of any periodontal treatment in the past 6 months
* patients with hormonal changes such as pregnancy or lactation; and 5) patients having fixed dentures or removable prothesis
* OSAS treatment started (using OSAS therapy device or undergoing surgical operation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Serum Total Antioxidant Status (TAS) level (millimolar per liter (mmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Serum Total Oxidant Status (TOS) level (mikromolar per liter (µmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Serum Oxidative Stress Index (OSI) level : TOS/TAS | 3 months
  Changes in serum and salivary oxidative stress parameters
Serum Native Thiol (mikromolar per liter (µmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Serum Thiol/disulfid (millimolar per liter (mmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Saliva Total Antioxidant Status (TAS) level (millimolar per liter (mmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Saliva Total Oxidant Status (TOS) level (mikromolar per liter (µmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Saliva Oxidative Stress Index (OSI) level : TOS/TAS | 3 months
  Changes in serum and salivary oxidative stress parameters
Saliva Native Thiol (mikromolar per liter (µmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters
Saliva Thiol/disulfid (millimolar per liter (mmol /L)) | 3 months
  Changes in serum and salivary oxidative stress parameters

SECONDARY OUTCOMES:
Plaque Index (PI) | 3 months
  Change in clinical measures of chronic periodontitis
Gingival Index (GI) | 3 months
  Change in clinical measures of chronic periodontitis
Bleeding on probing (BOP) | 3 months
  Change in clinical measures of chronic periodontitis
Clinical attachment loss(CAL) | 3 months
  Change in clinical measures of chronic periodontitis
Probing pocket depth (PD) | 3 months
  Change in clinical measures of chronic periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Betul Özsağır, Study Chair — Bezmialem VU
Locations (1):
- Bezmialem Vakıf University, Faculty of Dentistry, Deparment of Periodontology,, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loke W, Girvan T, Ingmundson P, Verrett R, Schoolfield J, Mealey BL. Investigating the association between obstructive sleep apnea and periodontitis. J Periodontol. 2015 Feb;86(2):232-43. doi: 10.1902/jop.2014.140229. Epub 2014 Oct 9. PMID 25299385
- [Result] Gamsiz-Isik H, Kiyan E, Bingol Z, Baser U, Ademoglu E, Yalcin F. Does Obstructive Sleep Apnea Increase the Risk for Periodontal Disease? A Case-Control Study. J Periodontol. 2017 May;88(5):443-449. doi: 10.1902/jop.2016.160365. Epub 2016 Nov 18. PMID 27858556
- [Result] DPTT study group; Engebretson S, Gelato M, Hyman L, Michalowicz BS, Schoenfeld E. Design features of the Diabetes and Periodontal Therapy Trial (DPTT): a multicenter randomized single-masked clinical trial testing the effect of nonsurgical periodontal therapy on glycosylated hemoglobin (HbA1c) levels in subjects with type 2 diabetes and chronic periodontitis. Contemp Clin Trials. 2013 Nov;36(2):515-26. doi: 10.1016/j.cct.2013.09.010. Epub 2013 Sep 27. PMID 24080100